CLINICAL TRIAL: NCT06370585
Title: Phase I Clinical Study to Evaluate the Safety and Tolerability of PRO-229 Ophthalmic Solution Compared to Lagricel® Ofteno PF in Clinically Healthy Subjects
Brief Title: Clinical Study to Evaluate the Safety and Tolerability of PRO-229 Ophthalmic Solution Compared to Lagricel® Ofteno PF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOPH229-0823/I
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — CD5L protein, human

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, comparative, double-masked, single-center, randomized, controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-229 (Experimental): * Dexpanthenol 2% and sodium hyaluronate 0.15% ophthalmic solution.
  * Dosage:1 drop QID [4] (four times per day) for 7 days on right both eyes.
  * Route of administration: Ophthalmic.
  * Presentation: Multidose dropper bottle.
  Interventions: Drug: PRO-229
- Lagricel® Ofteno PF (Active Comparator): * Sodium hyaluronate 0.4%. Ophthalmic solution.
  * Dosage: 1 drop QID [4] (four times per day) for 7 days on right both eyes.
  * Route of administration: Ophthalmic.
  * Presentation: Multidose dropper bottle.
  Interventions: Drug: Lagricel® Ofteno PF

INTERVENTIONS:
Drug: PRO-229 — - Dexpanthenol 2% and sodium hyaluronate 0.15% ophthalmic solution.
  Arms: PRO-229
Drug: Lagricel® Ofteno PF — - Sodium hyaluronate 0.4%. Ophthalmic solution.
  Arms: Lagricel® Ofteno PF

SUMMARY:
This is a phase I study evaluating safety and tolerability of PRO-229 ophthalmic solution through he incidence of unexpected adverse events, changes in Best Corrected Visual Acuity (BCVA), incidence of chemosis, and changes in ocular surface staining using the Sjögren's International Collaborative Clinical Alliance (SICCA) Ocular Staining Score (OSS) scale compared to Lagricel® Ofteno PF in clinically healthy subjects.

DETAILED DESCRIPTION:
The variables to be evaluated include:

Primary objective:

- To evaluate the safety and tolerability of PRO-229 ophthalmic solution compared to Lagricel® Ofteno PF in clinically healthy subjects.

Specific objective:

- To compare the safety of PRO-229 formulation compared to Lagricel® Ofteno PF through the incidence of adverse events related to both investigational products.

Secondary Objectives:

* To compare the safety of vs. PRO-229 formulation compared to Lagricel® Ofteno PF by changes in Best Corrected Visual Acuity (BCVA).
* To compare the safety of PRO-229 formulation compared to Lagricel® Ofteno PF by changes in ocular surface staining assessed with the the Sjögren's International Collaborative Clinical Alliance (SICCA) Ocular Staining Score (OSS) scale.
* To compare the safety of PRO-229 formulation compared to Lagricel® Ofteno PF by the incidence of chemosis.
* To compare the tolerability of PRO-229 formulation compared to Lagricel® Ofteno PF by changes in conjunctival hyperemia grades 3 or 4.
* To ompare the tolerability of PRO-229 formulation compared to Lagricel® Ofteno Ophthalmic PF by adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to voluntarily give their signed informed consent.
* Ophthalmologically and clinically healthy subjects.
* Being able to and willing to comply with scheduled visits, treatment plan, and other study procedures.
* Age between 18 to 45 years.
* Male or female gender.
* Women of childbearing potential who have not undergone Bilateral Tubal Occlusion (BTO [Tubal Ligation]), hysterectomy, or bilateral oophorectomy must ensure continuation (initiated ≥ 30 days prior to signing the informed consent form [ICF]) of the use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Best corrected visual acuity (BCVA) of 20/30 or better in both eyes.
* Corneal staining ≤ grade I on the Oxford Scale.
* Having an intraocular pressure ≥ 10 and ≤ 21 mmHg.

Exclusion Criteria:

* History of hypersensitivity to fluoroquinolones, steroid anti-inflammatories, or any of the components of the drugs under investigation.
* Use of ophthalmic medications from any pharmacological group.
* Use of medications by any other route of administration.
* Use of non-steroidal anti-inflammatory drugs, steroid anti-inflammatory drugs, or antibiotics by any route of administration in the last 30 days.
* History of eye surgery in the last 6 months.
* Use of contact lenses for a period less than two weeks prior to the start of the study, and during the intervention period of this study.
* In the case of women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Having participated in any clinical research study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* History of any chronic-degenerative disease, including Diabetes Mellitus or Systemic Arterial Hypertension.
* Diagnosis of glaucoma or ocular hypertension.
* Known diagnosis of liver or heart disease.
* Presenting active inflammatory or infectious disease at the time of entry into the study.
* Presenting unresolved lesions or traumas at the time of entry into the study.
* Having been subjected to non-ophthalmological surgical procedures in the last 3 months.
* Being or having an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is an employee of the research site or the sponsor, and who directly participates in this study.
* Active smoking (specified as the consumption of cigarettes regardless of the amount and frequency, 4 weeks prior to study inclusion and during the intervention period of this study).
* Active alcoholism (specified as the consumption of alcoholic beverages, regardless of the amount and frequency, 72 hours prior to study inclusion and during the intervention period of this study).

Elimination Criteria

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the compounds used during the tests -(fluorescein, tetracaine).
* Non-tolerability or hypersensitivity to any of the drugs under investigation.
* Adherence < 80% determined by the subject's diary and corroborated by the final weight of the research products (RP) compared to the initial weight.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence Unexpected Related Adverse Reactions | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), 3 (Visit 1), 8 (Final Visit) and 12 (Safety Call) after the inclusion of each subject.
  Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention.

SECONDARY OUTCOMES:
Changes in Best Corrected Visual Acuity (BCVA) | Through an average of 8 days. Evaluations will take place on days 0 (Basal Visit), 3 (Visit 1), and 8 (Final Visit) after the inclusion of each subject.
  BCVA will be evaluated through Snellen chart
Changes in ocular surface staining using SICCA ocular staining score scale | Through an average of 8 days. Evaluations will take place on days 0 (Basal Visit), 3 (Visit 1), and 8 (Final Visit) after the inclusion of each subject.
  Changes in ocular surface staining will be evaluated using the Sjögren's International Collaborative Clinical Alliance (SICCA) Ocular Staining Score (OSS) scale compared to Lagricel® Ofteno PF in clinically healthy subjects.
Incidence of chemosis | Through an average of 8 days. Evaluations will take place on days 0 (Basal Visit), 3 (Visit 1), and 8 (Final Visit) after the inclusion of each subject.
  Incidence of chemosis will be evaluated through direct observation by principal investigator
  0 = Absent
  1 = Present
Incidence of grade 3 or 4 conjunctival hyperemia. | Through an average of 8 days. Evaluations will take place on days 0 (Basal Visit), 3 (Visit 1), and 8 (Final Visit) after the inclusion of each subject.
  Conjunctival hyperemia will be evaluated through Efron grading scale.
Adherence to treatment (adherence) | Through an average of 8 days. This evaluations will take place on days 8 (Final Visit) after the inclusion of each subject.
  Adherence will be evaluated through the treatment record in the subject's diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion Mexicana para la Investigacion Clinica, Pachuca, Hidalgo, Mexico

IPD SHARING:
Plan to Share IPD: No